CLINICAL TRIAL: NCT04534439
Title: A Randomized, Placebo-controlled, Double-blinded, Multi-centre, Phase 2 Study to Assess Safety, Tolerability and Renal Effects of APX-115 in Subjects With Type 2 Diabetes and Nephropathy
Brief Title: Safety, Tolerability and Renal Effects of APX-115 in Subjects With Type 2 Diabetes and Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aptabio Therapeutics, Inc. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A01-115-02-EU; 2019-004155-37 (EudraCT Number)
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Nephropathies; Diabetes Mellitus, Type 2; Nephropathy, Diabetic
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — isuzinaxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APX-115 (Experimental): Oral administration of APX-115 400mg, daily
  Interventions: Drug: APX-115
- Placebo (Placebo Comparator): Oral administration of APX-115-matching placebo 400mg, daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APX-115 — oral administration of APX-115 400mg capsule once daily for 12 weeks
  Arms: APX-115
Drug: Placebo — oral administration of APX-115-matching placebo 400mg capsule once daily for 12 weeks
  Arms: Placebo

SUMMARY:
This is a proof of concept (PoC) trial to evaluate the safety, tolerability and renal effect of APX-115 in subjects with Type 2 diabetes and nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of type 2 diabetes and nephropathy
* First morning void (FMV) UACR between 200 and 3000 mg/g, inclusive
* 30 mL/min/1.73m2 ≤ eGFR ≤ 90 mL/min/1.73m2 using CKD-EPI formula at screening
* HbA1c ≤ 10% at screening visit
* Subject who has been taking unchanged dosage of ACE inhibitor or ARB medication for at least 3 months prior to screening and is not anticipated to change its dosage during the course of the study
* Willing to be under dietary management for diabetes

Exclusion Criteria:

* History of type 1 diabetes mellitus or gestational diabetes
* Subject's renal impairment and/or albuminuria is considered to be of origin other than Diabetic Kidney Disease
* Subject with uncontrolled blood pressure
* Clinically significant abnormal laboratory findings
* History of any cardiovascular event within 6 months prior to screening or cardiovascular procedure planned during the clinical trial
* Diagnostic or interventional procedure requiring a contrast agent within 4 weeks before the screening visit or planned during the course of the study
* Clinically significant ECG abnormalities on a 12-lead ECG at the screening visit or before randomization
* Current or history of NYHA class IV heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Mean change in urine albumin to creatinine ratio (UACR) in APX-115 group compared to placebo group | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Istavan Wittmann, MD, Principal Investigator — University of Pecs
Locations (16):
- Bulgaria (10):
  - Pleven, Pleven
  - Sveta Karidad, Plovdiv
  - Diagnostic-consultative centre I, Sliven
  - Hadzhi Dimitar, Sofia
  - HERA, Sofia
  - Medical center - Sveti Dimitar, Sofia
  - Sirtuin, Sofia
  - Sveta, Sofia
  - Hristo Botev, Vratsa
  - Sveti Panteleymon Yambol, Yambol
- Nefromed s.r.o, Prague, Czechia
- Hungary (3):
  - Drug Research Center, Balatonfüred
  - UNO MEDICAL Trials Kft., Budapest
  - Mint House Private Medical Center, Székesfehérvár
- Serbia (2):
  - Bezanijska Kosa, Belgrade
  - Clinical Centre of Serbia, clinic for endocrinology, diabetes and metabolism diseases, department for obesity, metabolic and reproductive disorders, Belgrade

IPD SHARING:
Plan to Share IPD: Undecided